CLINICAL TRIAL: NCT05454410
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Single Subcutaneous MIJ821 Injection in Addition to Standard of Care in Participants With Treatment-resistant Depression
Brief Title: Study of Efficacy, Safety, Tolerability and Pharmacokinetics of MIJ821 in Participants With Treatment- Resistant Depression (TRD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMIJ821B12201; 2021-005992-38 (EudraCT Number)
Record Dates: First submitted 2022-06-16; First posted 2022-07-12 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Treatment-Resistant Depression
Keywords: Treatment-Resistant Depression; Major Depressive Episode; Major Depressive Disorder; MIJ821; Anti-depressive Agent; Subcutaneous; Placebo; Adult
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MIJ821 1 mg (Experimental): Participants received a single dose of 1 mg MIJ821 administered as a subcutaneous (SC) injection on Day 1.
  Interventions: Drug: MIJ821 Subcutaneous Injection 1 mg
- MIJ821 4 mg (Experimental): Participants received a single dose of 4 mg MIJ821 administered as an SC injection on Day 1.
  Interventions: Drug: MIJ821 Subcutaneous Injection 4 mg
- MIJ821 10 mg (Experimental): Participants received a single dose of 10 mg MIJ821 administered as an SC injection on Day 1.
  Interventions: Drug: MIJ821 Subcutaneous Injection 10 mg
- Placebo (Placebo Comparator): Participants received a single dose of 0.9% sodium chloride solution administered as an SC injection on Day 1.
  Interventions: Drug: Placebo Subcutaneous Injection

INTERVENTIONS:
Drug: MIJ821 Subcutaneous Injection 1 mg — MIJ821 supplied in vials as a powder for solution for injection, reconstituted and administered as a single SC injection on Day 1.
  Arms: MIJ821 1 mg
Drug: MIJ821 Subcutaneous Injection 4 mg — MIJ821 supplied in vials as a powder for solution for injection, reconstituted and administered as a single SC injection on Day 1.
  Arms: MIJ821 4 mg
Drug: MIJ821 Subcutaneous Injection 10 mg — MIJ821 supplied in vials as a powder for solution for injection, reconstituted and administered as a single SC injection on Day 1.
  Arms: MIJ821 10 mg
Drug: Placebo Subcutaneous Injection — 0.9% sodium chloride solution administered as a single SC injection on Day 1.
  Arms: Placebo

SUMMARY:
The main purpose of this study was to evaluate safety and efficacy of a single injection of MIJ821 in addition to standard of care (SoC) pharmacological anti-depressant treatment in participants with treatment-resistant depression (TRD)

DETAILED DESCRIPTION:
The trial included a screening period of up to 28 days. On Day 1, after screening, eligible participants were randomized to one of the treatment arms (1 mg, 4 mg, or 10 mg of MIJ821) or placebo and received study treatment administered as a single subcutaneous injection. Participants remained at the clinic for at least 4 hours after administration of study treatment for safety observation including assessment of local tolerability by visual inspection of the injection area. Post-dose clinic visits occurred 24 hours post dose (Day 2), Days 8, 15, 22 and 29 to evaluate efficacy and safety. Efficacy assessments included the Montgomery-Asberg Depression Scale (MADRS) and other clinical outcome assessments (COAs). Safety assessments included laboratory tests, ECGs, vital signs and physical examinations. In addition, phone calls were conducted 3 days after each on-site clinic visit with the exception of the End-of-study (EOS) visit. EOS visit was completed on site on Day 29. Including screening, participants were in the study for up to 8 weeks (57 days).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to participation in the study
* Male and female participants, 18 to 65 years of age (inclusive) at screening
* DSM-5 defined major depressive disorder (MDD) and a current major depressive episode (MDE)
* MADRS score ≥ 24
* Failure to respond to 2 or more antidepressant treatments where the two failed treatments are two different antidepressants

Exclusion Criteria:

* Any prior or current diagnosis of MDD with psychotic features, bipolar disorder, schizophrenia, or schizoaffective disorder
* Participants with acute alcohol or substance use disorder or withdrawal symptoms requiring detoxification, or participants who went through detoxification treatment within 1 month before Screening
* Participants with current borderline personality disorder or antisocial personality disorder
* Current clinical diagnosis of autism, dementia, or intellectual disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (3):
  - 25Uni of Alabama at Birmingham, Birmingham, Alabama
  - Research Centers of America LLC, Oakland Park, Florida
  - Interventional Psychiatry Tampa Bay, Tampa, Florida
- Japan (3):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Swiecie North West
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Boi de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All inclusion and exclusion criteria were checked during screening and on Day 1, prior to randomization.
Groups:
- MIJ821 10 mg: Participants received a single dose of 10 mg MIJ821 administered as a subcutaneous (SC) injection on Day 1.
- MIJ821 4 mg: Participants received a single dose of 4 mg MIJ821 administered as a SC injection on Day 1.
- MIJ821 1 mg: Participants received a single dose of 1 mg MIJ821 administered as a SC injection on Day 1.
- Placebo: Participants received a single dose of 0.9% sodium chloride solution administered as a SC injection on Day 1.
Period: Overall Study
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo
Started | 15 | 14 | 14 | 17
Completed | 15 | 14 | 13 | 16
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized set included all Randomized participants.
Groups:
- MIJ821 10 mg: Participants received a single dose of 10 mg MIJ821 administered as a subcutaneous injection on Day 1.
- MIJ821 4 mg: Participants received a single dose of 4 mg MIJ821 administered as a subcutaneous injection on Day 1.
- MIJ821 1 mg: Participants received a single dose of 1 mg MIJ821 administered as a subcutaneous injection on Day 1.
- Placebo: Participants received a single dose of 0.9% sodium chloride solution administered as a subcutaneous injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 14 | 17 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.36) | 43.9 (11.29) | 46.9 (9.73) | 47.1 (12.05) | 46.5 (11.26)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 4 | 5 | 10 | 23
  Female | 11 | 10 | 9 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 0 | 8
  Not Hispanic or Latino | 13 | 11 | 11 | 17 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 13 | 12 | 17 | 57
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian / Japanese | 0 | 1 | 2 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score 24 Hours (Day 2) After Injection
Description: The Montgomery Åsberg Depression Rating Scale (MADRS, SIGMA version), is a clinician rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 0 - 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts and suicidal thoughts. The MADRS scores were collected electronically by qualified personnel.
Time Frame: Baseline and 24 hours after SC injection
Population: The Full Analysis Set (FAS) included all randomized participants who received a dose of the randomized treatment. Participants were analyzed according to the assigned treatment groups.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Groups:
- MIJ821 10 mg: Participants received a single dose of 10mg MIJ821 administered as a subcutaneous (SC) injection on Day 1.
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 17
Scores on a Scale | -14.1 (1.95) | -11.4 (2.04) | -8.4 (2.02) | -8.9 (1.82)
Statistical Analysis 1: Comparison: MIJ821 10 mg vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Net) = -5.2, 90% CI 2-sided [-9.6 to -0.7] — Placebo adjusted means (MIJ821-Placebo). 90% CIs are nominal and not adjusted for multiplicity
Statistical Analysis 2: Comparison: MIJ821 4 mg vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Net) = -2.5, 90% CI 2-sided [-7.0 to 2.1] — Placebo adjusted means (MIJ821-Placebo). 90% CIs are nominal and not adjusted for multiplicity
Statistical Analysis 3: Comparison: MIJ821 1 mg vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Net) = 0.6, 90% CI 2-sided [-4.0 to 5.1] — Placebo adjusted means (MIJ821-Placebo). 90% CIs are nominal and not adjusted for multiplicity

2. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs), Including Adverse Events of Special Interest (AESIs)
Description: A TEAE was defined as an adverse event starting or worsening after the administration of study medication and up to the end of study visit. The following events were considered AESIs:
  * Dissociation
  * Sedation
  * Cardiovascular effects (Blood Pressure changes and QT interval prolongation on electrocardiogram [ECG])
  * Respiratory effects (difficulty in breathing, changes in oxygen saturation)
  * Suicidality (suicidal ideation or behavior)
  * Memory gaps/amnesia
  * Cystitis or lower urinary tract adverse events
Time Frame: From Day 1 after SC injection to end of study, up to 29 Days
Population: The Safety Analysis Set included all participants who received any study drug. Participants were analyzed according to the study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 17
Participants
  With at least one AE | 10 | 6 | 4 | 7
  With at least one AESI | 9 | 5 | 2 | 3
  Blood pressure increased | 0 | 1 | 1 | 0
  Dissociation | 5 | 2 | 0 | 2
  Derealization | 1 | 0 | 0 | 0
  Vision blurred | 0 | 0 | 1 | 0
  Amnesia | 1 | 0 | 0 | 0
  Somnolence | 4 | 1 | 0 | 1
  Sedation | 1 | 1 | 0 | 0

3. Secondary Outcome: Pharmacokinetics (PK) of MIJ821 in Plasma for Area Under the Curve From the Time of Dosing to the Time of the Last Measurable Concentration (AUClast)
Description: Blood samples were collected at the indicated time points for PK analysis. AUClast was defined as the area under the curve from time zero to the last measurable concentration sampling time (tlast).
Time Frame: Baseline, 0.17 hour, 0.33 hour, 0.5 hour, 0.75 hour, 1, 1.5, 2, 4 and 24 hours post injection
Population: The PK analysis set included all participants with at least one available, valid PK concentration measurement, who received any study drug and with no protocol deviations that had an impact on PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg
Number analyzed (Participants) | 15 | 13 | 13
h*ng/mL | 231 (33.5) | 89.5 (45.7) | 5.92 (85.1)

4. Secondary Outcome: PK of MIJ821 in Plasma for Maximum Serum Concentration (Cmax)
Description: Blood samples were collected at the indicated time points for PK analysis. Cmax was defined as the maximum (peak) observed plasma drug concentration after single dose administration.
Time Frame: Baseline, 0.17 hour, 0.33 hour, 0.5 hour, 0.75 hour, 1, 1.5, 2, 4 and 24 hours post injection
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg
Number analyzed (Participants) | 15 | 13 | 13
ng/mL | 42.7 (37.2) | 17.5 (46.7) | 2.32 (55.4)

5. Secondary Outcome: PK of MIJ821 in Plasma for Time to Maximum Drug Concentration (Tmax)
Description: Blood samples were collected at the indicated time points for PK analysis. Tmax was defined as the time to reach maximum (peak) plasma drug concentration after single dose administration (time).
Time Frame: Baseline, 0.17 hour, 0.33 hour, 0.5 hour, 0.75 hour, 1, 1.5, 2, 4 and 24 hours post injection
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (h)
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg
Number analyzed (Participants) | 15 | 14 | 14
hour (h) | 0.750 [0.333 to 2.00] | 0.500 [0.150 to 1.00] | 0.500 [0.167 to 0.783]

6. Secondary Outcome: Change From Baseline in the MADRS Total Scores at Day 8, 15, 22 and 29 Visits
Description: The MADRS (SIGMA version), is a clinician rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 0 - 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts and suicidal thoughts. The MADRS scores were collected electronically by qualified personnel.
Time Frame: Baseline, Days 8, 15, 22 and 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 17
Scores on a Scale
  Change from Baseline (Day 8) | -15.3 (2.0) | -9.9 (2.1) | -8.2 (2.0) | -7.4 (1.8)
  Change from Baseline (Day 15): number analyzed (Participants) | 14 | 13 | 14 | 17
  Change from Baseline (Day 15) | -14.0 (2.2) | -8.5 (2.2) | -11.0 (2.2) | -7.7 (2.0)
  Change from Baseline (Day 22): number analyzed (Participants) | 14 | 14 | 13 | 17
  Change from Baseline (Day 22) | -14.9 (2.2) | -10.7 (2.3) | -9.7 (2.3) | -7.0 (2.0)
  Change from Baseline (Day 29): number analyzed (Participants) | 14 | 14 | 13 | 16
  Change from Baseline (Day 29) | -14.9 (2.3) | -12.7 (2.4) | -10.7 (2.4) | -7.0 (2.1)

7. Secondary Outcome: Dose-response (DR) Relationship of MIJ821 With Respect to Change From Baseline in MADRS Total Score at 24 Hours After Single SC Injection
Description: The multiple comparison procedure - modelling (MCP-Mod) approach was an integrated approach used to investigate DR relationships, while confirming efficacy of the test product based on hypothesis testing. A set of candidate models was tested using Multiple Comparison Procedures (MCP) that preserve the family-wise error rate (FWER) to determine the model best representing the underlying DR. Efficacy via DR was established when at least one of the model tests was signiﬁcant.
Time Frame: Baseline up to 24 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 10 mg | MIJ821 4 mg | MIJ821 1 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 17
Scores on a Scale | -14.1 (1.95) | -11.4 (2.04) | -8.4 (2.02) | -8.9 (1.82)
Statistical Analysis 1: Comparison: MIJ821 10 mg vs MIJ821 4 mg vs MIJ821 1 mg vs Placebo; MCP-Mod was used to check if there was a DR relationship between the change from baseline to 24 hours in MADRS total score and the doses received. The Least squares means under the primary estimand were used to test the null hypothesis of a flat DR relationship at a one-sided significance level of 5% against the alternative hypothesis of a non-flat DR curve. Six candidate DR curves were used to derive the optimal model contrasts for the multiple contrast tests. A monotone DR was assumed; Test type: Superiority; p = 0.0242, Multiple contrast test — P-value for the selected model best representing the underlying DR (the lowest p-value out of the 6 candidate models), adjusted for multiple comparisons

8. Secondary Outcome: Exposure-response Relationship of MIJ821 With Respect to Change From Baseline in MADRS Total Score. Estimated Parameters: Placebo Effect E0, Emax
Description: The exposure-response relationship was investigated considering PK exposure parameters (AUClast and Cmax) and the change from baseline MADRS score derived at 4 h and 24 h after injection and Day 8, Day 15, Day 22 and Day 29 during the follow-up.
  The emax model or sigmoid emax model were planned to be fitted for the change from baseline at each follow up visit and the PK exposure parameters, Cmax and AUClast. If the model converges, parameters estimated from the Sigmoid emax model are: the placebo effect E0, EC50, Emax and the hill parameter.
Time Frame: Baseline, Day 2, 15, 22 and 29
Population: as for outcome 3
Measure: Number; unit: Scores on a scale
Groups:
- Overall: Pooled for all participants
Arm/Group | Overall
Number analyzed (Participants) | 41
Scores on a scale
  Exposure-response Relationship Cmax: placebo effect E0 | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues
  Exposure-response Relationship Cmax: Emax | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues
  Exposure-response Relationship AUClast: placebo effect E0 | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues
  Exposure-response Relationship AUClast: Emax | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues

9. Secondary Outcome: Exposure-response Relationship of MIJ821 With Respect to Change From Baseline in MADRS Total Score. Estimated Parameter: EC50 (Cmax)
Description: as for outcome 8
Time Frame: Baseline, Day 2, 15, 22 and 29
Population: as for outcome 3
Measure: Number; unit: ng/mL
Arm/Group | Overall
Number analyzed (Participants) | 41
ng/mL | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues

10. Secondary Outcome: Exposure-response Relationship of MIJ821 With Respect to Change From Baseline in MADRS Total Score. Estimated Parameter: EC50 (AUClast)
Description: as for outcome 8
Time Frame: Baseline, Day 2, 15, 22 and 29
Population: as for outcome 3
Measure: Number; unit: h*ng/mL
Arm/Group | Overall
Number analyzed (Participants) | 41
h*ng/mL | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues

11. Secondary Outcome: Exposure-response Relationship of MIJ821 With Respect to Change From Baseline in MADRS Total Score. Estimated Parameter: Hill Parameter
Description: as for outcome 8
Time Frame: Baseline, Day 2, 15, 22 and 29
Population: as for outcome 3
Measure: Number; unit: Hill coefficient
Arm/Group | Overall
Number analyzed (Participants) | 41
Hill coefficient
  Exposure-response Relationship Cmax: Hill parameter | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues
  Exposure-response Relationship AUClast: Hill parameter | NA — estimates in the Sigmoid emax (or Emax) model were not available due to non-convergence issues

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, up to a maximum duration of 29 days.
Description: The Safety Analysis Set included all participants who received any study drug. Participants were analyzed according to the study treatment received.
Groups:
- MIJ821 4mg: Participants received a single dose of 4 mg MIJ821 administered as a SC injection on Day 1.
- MIJ821 1mg: Participants received a single dose of 1 mg MIJ821 administered as a SC injection on Day 1.
- All MIJ821: All MIJ821 Dosages
- All Participants: All Participants included in the Safety Analysis Set
Arm/Group | MIJ821 10 mg | MIJ821 4mg | MIJ821 1mg | Placebo | All MIJ821 | All Participants
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/17 | 0/43 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/17 | 0/43 | 0/60
Other Adverse Events (participants affected / at risk) | 10/15 | 6/14 | 4/14 | 7/17 | 20/43 | 27/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIJ821 10 mg (N=15) | MIJ821 4mg (N=14) | MIJ821 1mg (N=14) | Placebo (N=17) | All MIJ821 (N=43) | All Participants (N=60)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Injection site erythema (General disorders) | 3 | 0 | 0 | 0 | 3 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 2
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 3 | 0 | 1 | 3 | 4 | 7
Sedation (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 2
Somnolence (Nervous system disorders) | 4 | 1 | 0 | 1 | 5 | 6
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1
Derealisation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dissociation (Psychiatric disorders) | 5 | 2 | 0 | 2 | 7 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT05454410/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05454410/SAP_001.pdf